CLINICAL TRIAL: NCT03203811
Title: A Phase 1, Double-blind, Placebo-Controlled, Single Oral Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HTI-2088 Tablet in Healthy Adult Subjects
Brief Title: A Phase 1, Study to Evaluate HTI-2088 Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hengrui Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTI-2088-101
Record Dates: First submitted 2017-06-12; First posted 2017-06-29 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diabetes
Keywords: Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): 2mg, HTI-2088 oral tablet or placebo, one dose, evaluate over 4 days
  Interventions: Drug: HTI-2088; Drug: Placebo
- Middle Dose (Experimental): 3.75mg HTI-2088 oral tablet or placebo, one dose, evaluate over 4 days
  Interventions: Drug: HTI-2088; Drug: Placebo
- High Dose (Experimental): 5mg HTI-2088 oral tablet or placebo, one dose, evaluate over 4 days
  Interventions: Drug: HTI-2088; Drug: Placebo

INTERVENTIONS:
Drug: HTI-2088 — 3 dose levels
Drug: Placebo — placebo oral tablet

SUMMARY:
Single Center, Randomized, Double Blind, Placebo Controlled, Single ascending dose trial at 3 levels. Ten subjects will be enrolled at each dose.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, single ascending dose trial with single oral doses of HTI-2088 tablets to subjects at 3 levels (2.5, 3.75, 5 mg). Ten subjects will be enrolled at each dose level, randomized within groups at an active: placebo ratio of 4:1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18 and 55 years of age (inclusive), without diabetes FPG <126 mg/dL.
2. Body mass index (BMI) of 19 to 30 kg/m2 (inclusive); and a total body weight ≥50 kg.
3. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. An informed consent document signed and dated by the subject.
5. Male subjects must agree to utilize a highly effective method of contraception (condom with or without spermicide) during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 90 days following IP dosing, and must agree to refrain from sperm donation from Day 0 until at least 90 days after the IP dose.
6. Females must meet at least one of the following criteria:

   * sexually inactive (abstinent) for at least 14 days prior to the first dose, throughout the study and for 90 days after IP dose
   * postmenopausal, defined by at least 12 consecutive months of amenorrhea without an alternative medical cause
   * using one of the following acceptable birth control methods: surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to the first dose; intra-uterine device in place for at least 3 months prior to the first dose; barrier method (condom, diaphragm) with spermicide for at least 14 days prior to the first dose, throughout the study and for 90 days after IP dose; surgical sterilization of the partner (vasectomy for at least 6 months prior to the first dose); hormonal contraception for at least 3 months prior to the first dose, throughout the study and for 90 days after IP dose.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or drug allergies. In particular, any history or evidence at Screening of chronic GI disorders (e.g., celiac sprue, ulcerative colitis, Crohn's disease, etc.), thyroid disease, or pancreatitis, any condition possibly affecting drug absorption (e.g., gastrectomy).
2. History of gastrointestinal surgery within one year of the screening visit.
3. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that could have increased the risk associated with study participation or investigational product administration or could have interfered with the interpretation of study results and, in the judgment of the investigator, made the subject inappropriate for entry into the study.
4. Positive results of alcohol or substances of abuse at screening or upon admission to the clinical research unit.
5. A positive pregnancy test at screening and upon admission to the clinical research unit, or subject is lactating, if the subject is female.
6. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounce (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening; Consumption of alcohol within 24 hours of receiving IP.
7. Treatment with any investigational drug within 30 days or 5 half-lives preceding the first dose of IP.
8. Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study.
9. Blood donation of approximately 1 pint (approximately 473 mL) or more within 56 days, or plasma donation within 7 days of receiving IP.
10. Use of prescription, nonprescription drugs, illicit drug use, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of IP. Herbal supplements and hormone replacement therapy should be discontinued 28 days prior to the first dose of IP.
11. Evidence of human immunodeficiency virus (HIV)/ hepatitis C/ hepatitis B infection and/or positive human HIV/hepatitis C/hepatitis B antibodies (a negative test result within the 3 months prior to screening may be used instead of obtaining a screening laboratory sample for these laboratory tests)
12. History of using GLP-1 analogs.
13. Known sensitivity to any of the components of the investigational product formulation or SNAC
14. Current smoker or user of any tobacco products.
15. Consumption of any grapefruit or grapefruit-containing juices within 14 days of receiving the IP.
16. Consumption of any caffeine- or xanthine-containing foods or beverages within 24 hours of receiving IP.
17. Have poor venous access and are unable to donate blood.
18. In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.
19. Subjects who are investigational site staff members or subjects who are Sponsor employees directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1 week
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Cmax | 1 week
  Peak Plasma Concentration (Cmax)
AUC | 1 Week
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
PD Effects | 1 week
  effects on Glucose, Insulin, Insulin C-peptide
Glucose | 1 week
  Number of patients with effects on Glucose, Insulin, Insulin C-peptide
Insulin | 1 week
  Number of patients with effects on Insulin and Insulin C-peptide

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No